CLINICAL TRIAL: NCT02233842
Title: Cognitive Testing of Tobacco Use Measurement Items for Administration With Cancer Patients and Survivors
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Stephanie Land, Ph.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140189; 14-C-0189
Record Dates: First submitted 2014-09-06; First posted 2014-09-09 (Estimated); Results first posted 2016-07-27 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-08

CONDITIONS: Lung Cancer; Prostate Cancer; Bladder Cancer; Thymic Cancer
Keywords: Qualitative Data; Questionnaire
MeSH Terms: conditions — Lung Neoplasms; Prostatic Neoplasms; Urinary Bladder Neoplasms; Thymus Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tobacco Use in Cancer Pts & Survivors: Cognitive testing (e.g. participant interview) of tobacco use in patients (pts) who have cancer and who have survived cancer.
  Interventions: Behavioral: Participant interview

INTERVENTIONS:
Behavioral: Participant interview — People with cancer and who have survived cancer will have a 1 hour interview about using cigarettes and other tobacco products.

SUMMARY:
Background:

- People who have cancer have more medical problems if they smoke. Some studies show that smoking even makes cancer treatment less effective. Researchers want to teach people about how tobacco use affects people after a cancer diagnosis. They want to come up with questions for people who have cancer and who have survived cancer. The questions will be about using cigarettes and other tobacco products and about second-hand smoke.

The questions will be used to understand how using tobacco affects people with cancer before, during, and after treatment. This will help doctors plan how to treat people with cancer and create programs to help people quit smoking in the future.

Objective:

- To evaluate and refine questions that assess tobacco use.

Eligibility:

- Adults age 21 or older who have cancer or are cancer survivors. The cancer can be at any site and any stage.

Design:

* This study will take about 1 hour.
* Participants will meet one-on-one with an interviewer. They will fill out a questionnaire and talk about the questions. Participants will explain how easy or hard it was to answer the questions and how they decided on their answers.
* All participants will be asked the same or very similar questions. Specific questions will be based on the participants own experiences with tobacco products.
* There will be no follow-up activities.

DETAILED DESCRIPTION:
Background:

Studies comparing cancer patients who smoke cigarettes at the time of diagnosis to former or never smokers have demonstrated increased difficulty with surgical wound healing and more treatment morbidity; reduced radiation and chemotherapy efficacy; reduced time to recurrence, progression, and second primary cancers; and increased mortality. Some studies have found that smoking interacts with cancer therapy efficacy.

Cigarette smoking is prevalent among patients with lung and head and neck cancers, with rates as high as 40% to 60% as of the time of diagnosis. The rate of smoking among cancer survivors has been estimated as 21% for lung cancer survivors and 39% for survivors of other cancers.(11)

Only 22% of NCI-funded phase III trials conducted by Cooperative Groups record patients cigarette smoking status among patients at the time of enrollment, and 4% record cigarette smoking status during follow-up.

We need to examine the impact of tobacco use on a wider range of therapeutic regimens and settings, with more detailed longitudinal tobacco use assessment. Research in this area is impeded by inadequate assessment of tobacco use after cancer diagnosis and a lack of valid, harmonized measures that are tailored to the trajectory of cancer diagnosis, treatment and survivorship.(15) The NCI-AACR Cancer Patient Tobacco Use Assessment Task Force formed in 2013 to develop recommendations for assessing tobacco use by cancer patients. The long- range goal of the Task Force is to advance the state of knowledge about the effect of tobacco use after a cancer diagnosis, to inform cancer treatment decision-making and to guide patients and providers regarding the timing and clinical significance of tobacco cessation.

Objectives:

To evaluate and refine proposed questionnaire items that assess tobacco use.

Eligibility:

Cancer patients with any disease site, stage, and extent of prior therapy and age greater than or equal to 21 years.

Design:

This study will evaluate and refine proposed questionnaire items that assess tobacco use in the cancer patient and survivor population. This study is purely qualitative. No research hypotheses will be tested in this study. There will be no therapy, administration of agent(s), or imaging administered as part of this study. Participants will only be asked to answer questions and then discuss their answers to the questions.

Patients who consent will participate in a session that will last up to one hour. They will complete a questionnaire about tobacco use and answer debriefing questions so that the interviewer can assess question comprehension, ease of answering, and accuracy of response.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with any prior confirmed cancer diagnosis being treated or followed at the Center for Cancer Research, Bethesda, Maryland, will be eligible.

3.1.1 Cancer patients with any disease site, stage, and extent of prior therapy will be eligible.

3.1.2 Patients age 21 years old and over will be eligible. The items are intended for use with an adult population, so we need to test with representatives of that population.

3.1.3 Additional eligibility criteria:

* Individuals must be able to understand and willing to answer items about their own tobacco use.
* Individuals must be able to read and speak English. For purposes of this study, we will limit participation to adults who can self-consent and self-report in English (vs. only being able to respond with the aid of a translator). The materials have been developed in English; this is intended to be cognitive testing of an English language questionnaire. (If a Spanish translation of the items will be developed in the future, a separate cognitive testing effort will be needed to ensure cultural equivalence of the items.)

3.1.4 Participants must be able to understand and be willing to sign a written informed consent

document. All participants will be asked to provide explicit consent.

3.1.5 Participants are eligible whether they have never used tobacco products of any type, used any type of tobacco previously, or are current tobacco users of any type. (Participant recruitment will be designed to enroll a variety of patients with respect to tobacco use.)

EXCLUSION CRITERIA:

None. (Patients may have already begun protocol treatment.)

INCLUSION OF WOMEN AND MINORITIES:

Both men and women of all races and ethnic groups are eligible for participation in testing of the items. In fact, to the extent possible, we will try to include diversity of demographic characteristics (age, race, gender, education level).

Ages: 21 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 21 or older who have cancer or are cancer survivors. The cancer can be at any site and any stage.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie R. Land, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Land SR, Warren GW, Crafts JL, Hatsukami DK, Ostroff JS, Willis GB, Chollette VY, Mitchell SA, Folz JN, Gulley JL, Szabo E, Brandon TH, Duffy SA, Toll BA. Cognitive testing of tobacco use items for administration to patients with cancer and cancer survivors in clinical research. Cancer. 2016 Jun 1;122(11):1728-34. doi: 10.1002/cncr.29964. Epub 2016 Mar 28. PMID 27019325
- [Result] Land SR, Toll BA, Moinpour CM, Mitchell SA, Ostroff JS, Hatsukami DK, Duffy SA, Gritz ER, Rigotti NA, Brandon TH, Prindiville SA, Sarna LP, Schnoll RA, Herbst RS, Cinciripini PM, Leischow SJ, Dresler CM, Fiore MC, Warren GW. Research Priorities, Measures, and Recommendations for Assessment of Tobacco Use in Clinical Cancer Research. Clin Cancer Res. 2016 Apr 15;22(8):1907-13. doi: 10.1158/1078-0432.CCR-16-0104. Epub 2016 Feb 17. PMID 26888828
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-C-0189.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Thirty-five subjects were recruited for this trial but three were unavailable due to time constraints, one was hesitant to participate and one refused to participate. As a result, only 30 subjects were enrolled in the trial. Five participants were assessed for each of the 6 different questionnaires to total 30 participants.
Groups:
- Tobacco Use in Cancer Patients and Survivors: Cognitive testing (e.g. participant interview) of tobacco use in patients who have cancer and who have survived cancer.
  Participant interview: People with cancer and who have survived cancer will have a 1 hour interview about using cigarettes and other tobacco products.
  Three iterative rounds of testing of 10 patients each were planned in the protocol for revision and retesting.
Period: Questionnaire 1 Version 1
Arm/Group | Tobacco Use in Cancer Patients and Survivors
Started | 5
Completed | 5
Not Completed | 0
Period: Questionnaire 1 Version 2
Arm/Group | Tobacco Use in Cancer Patients and Survivors
Started | 5
Completed | 5
Not Completed | 0
Period: Questionnaire 2 Version 1
Arm/Group | Tobacco Use in Cancer Patients and Survivors
Started | 5
Completed | 5
Not Completed | 0
Period: Questionnaire 2 Version 2
Arm/Group | Tobacco Use in Cancer Patients and Survivors
Started | 5
Completed | 5
Not Completed | 0
Period: Questionnaire 3 Version 1
Arm/Group | Tobacco Use in Cancer Patients and Survivors
Started | 5
Completed | 5
Not Completed | 0
Period: Questionnaire 3 Version 2
Arm/Group | Tobacco Use in Cancer Patients and Survivors
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Cognitive testing (e.g. participant interview) of tobacco use in patients who have cancer and who have survived cancer.
  Participant interview: People with cancer and who have survived cancer will have a 1 hour interview about using cigarettes and other tobacco products
Arm/Group | All Participants
Number analyzed (Participants) | 30
Age, Customized [Number; unit: participants]
  Age 20-29 | 1
  Age 30-39 | 0
  Age 40-49 | 1
  Age 50-59 | 13
  Age 60-69 | 8
  Age 70-79 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 25
  Black | 4
  Asian/PI (Pacific Islander) | 1
Region of Enrollment [Number; unit: participants]
  United States | 30
Education (highest level completed) [Number; unit: participants]
  High School/GED | 7
  Some college | 11
  College degree | 4
  Postgraduate degree | 8
Cigarette smoking status [Number; unit: participants]
  Former (quit at least 1yr prior to diagnosis) | 17
  Former at enrollment;current at diagnosis | 6
  Current | 6
  Never (current cigar smoker) | 1
Diagnosis [Number; unit: participants]
  Prostate cancer | 9
  Bladder cancer | 3
  Lung cancer | 8
  Pancreatic cancer | 1
  Testicular cancer | 1
  Thyroid cancer | 1
  Pleural mesothelioma | 3
  Thymus cancer | 4
Type of Trials Participants Were Enrolled [Number; unit: participants]
  Tumor-directed therapy clinical trial | 21
  Observational study | 6
  Patients being screened for trial eligibility | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants to Achieve Saturation in an English-language Paper Questionnaire
Description: Saturation is defined as satisfactory measurement of performance without need of further review.
Time Frame: Last subject interviewed, an average of 5 months
Measure: Number; unit: participants
Groups:
- All Participants: People who have cancer and who have survived cancer
  Participant interview: People with cancer and who have survived cancer will have a 1 hour interview about using cigarettes and other tobacco products.
Arm/Group | All Participants
Number analyzed (Participants) | 30
participants | 30

2. Primary Outcome: Number of Smokers at the Time of the Interview
Description: Current, former, and cigar smokers at the time the interview (e.g. Cancer Patient Tobacco Use Questionnaire (C-TUQ)) was initiated.
Time Frame: Day 1 of interview
Measure: Number; unit: participants
Groups:
- All Participants: Cognitive testing (e.g. participant interview) of tobacco use in patients who have cancer and who have survived cancer.
  Participant interview: People with cancer and who have survived cancer will have a 1 hour interview about using cigarettes and other tobacco products.
  Three iterative rounds of testing of 10 patients each were planned in the protocol for revision and retesting.
Arm/Group | All Participants
Number analyzed (Participants) | 30
participants
  Current Smoker | 6
  Former Smoker (quit 4-54 years ago) | 23
  Cigar Smoker (never smoked cigarettes) | 1

3. Primary Outcome: Number of Current and Former Smokers Who Smoked Cigarettes at the Time of Their Cancer Diagnosis
Description: Current and former smokers who were smoking at the time of their cancer diagnosis.
Time Frame: Day 1 of interview
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 30
participants
  Current Smoker | 6
  Former Smoker | 6

4. Primary Outcome: Time From Cancer Diagnosis to the Date of the Interview
Description: Patients diagnosed with cancer who participated in the Cancer Patient Tobacco Use Questionnaire (C-TUQ).
Time Frame: up to 24 years
Measure: Median (Full Range); unit: years
Arm/Group | All Participants
Number analyzed (Participants) | 30
years | 3 [1 to 24]

ADVERSE EVENTS:
Groups:
- Tobacco Use in Cancer Patients and Survivors: People who have cancer and who have survived cancer
  Participant interview: People with cancer and who have survived cancer will have a 1 hour interview about using cigarettes and other tobacco products.
Arm/Group | Tobacco Use in Cancer Patients and Survivors
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No